CLINICAL TRIAL: NCT06512844
Title: The Efficacy of Mindfulness Based Intervention for the Management of Psychosocial Factors Associated With Emotional Intelligence in Adolescents With Physical Disability: a Randomized Control Trial
Brief Title: MBSR for Improving Emotional Intelligence in Adolescents With Physical Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Aleeza Sohail, Mphil Research Student, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AleezaUW
Record Dates: First submitted 2024-06-29; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Physical Disability
Keywords: emotional intelligence; mindfulness; physical disability
MeSH Terms: interventions — Mindfulness-Based Stress Reduction; Methods

STUDY DESIGN:
Intervention Model Description: This clinical trial aims to evaluate the effectiveness of a mindfulness-based intervention (MBI) in managing psychosocial factors associated with emotional intelligence (EI) in adolescents with physical disabilities. It also seeks to assess the safety and overall impact of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Participants who were assigned to interventional group were exposed to Urdu adapted and translated mindfulness-based stress reduction training. These participants received 8 weeks of intervention.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR) Intervention
- Control/Wait list Group (No Intervention): Participant who were assigned to Control Group did not receive any Intervention although they just received some relaxation breathing exercises.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) Intervention — The MBSR training program consist of 8-week group session with the duration of 45-60 minutes each. Participants of the experimental group were given Mindfulness based stress reduction intervention in which they practice different mindfulness techniques. Each week focused on motor, cognitive and emotional issues of students with physically disabled. All the techniques also included psycho education
  Arms: Interventional Group

SUMMARY:
This study aims to provide evidence on the effectiveness of mindfulness-based interventions in enhancing emotional intelligence and managing psychosocial challenges in adolescents with physical disabilities, potentially offering a valuable tool for improving their overall well-being.

Does the mindfulness-based intervention improve emotional intelligence in adolescents with physical disabilities? Does the psychosocial factors like psychological distress, self-compassion improve during the intervention? Are there any adverse effects associated with the mindfulness-based intervention? Researcher will give intervention and compare the control and experimental group in Time 1 and Time 2 respectively

DETAILED DESCRIPTION:
Title: The Efficacy of Mindfulness-Based Intervention for the Management of Psychosocial Factors Associated with Emotional Intelligence in Adolescents with Physical Disability: A Randomized Control Trial

Objective: This clinical trial aims to evaluate the effectiveness of a mindfulness-based intervention (MBI) in managing psychosocial factors associated with emotional intelligence (EI) in adolescents with physical disabilities. It also seeks to assess the safety and overall impact of the intervention.

Main Questions:

Does the mindfulness-based intervention improve emotional intelligence in adolescents with physical disabilities? Does the psychosocial factors like psychological distress, self-compassion improve during the intervention? Are there any adverse effects associated with the mindfulness-based intervention?

Study Design:

Participants: Adolescents aged 10-18 years with a diagnosed physical disability.

Intervention: Mindfulness-based intervention (MBI) compared to a control group receiving no intervention.

Duration: 8 weeks Follow-Up: Participants will be assessed at baseline, mid-intervention (4 weeks), immediately post-intervention (8 weeks), and at a 3-month follow-up.

Methodology:

Participants will be randomly assigned to one of two groups:

Intervention Group: Will participate in the mindfulness-based intervention, which includes weekly mindfulness sessions and daily mindfulness practices at home.

Control Group: Will not receive any intervention but will continue with their usual activities along with some breathing exercises by the researcher.

Procedures:

Mindfulness Sessions: Weekly group sessions led by a trained mindfulness instructor, focusing on techniques such as meditation, breathing exercises, and body awareness.

Daily Practice: Participants in the intervention group will be instructed to practice mindfulness techniques daily and will receive support materials (e.g., audio recordings, practice guides).

Assessment:

Emotional Intelligence: Measured using the Schulte Self-Report Emotional Intelligence Test (SSEIT) at all assessment points.

Psychosocial Factors: Evaluated using standardized questionnaires such as the Child and Adolescent Trauma Screen (CATS) and the Depression, Anxiety, and Stress Scales (DASS).

Adverse Effects: Monitored through regular check-ins and a diary where participants can record any negative experiences.

Visit Schedule:

Baseline Visit: Initial assessment and randomization. Weekly Check-ins: Short visits or calls to monitor progress and adherence. Mid-Intervention (4 weeks): Comprehensive assessment of EI and psychosocial factors.

Post-Intervention (8 weeks): Final assessment of EI and psychosocial factors, collection of feedback on the intervention.

3-Month Follow-Up: Long-term assessment of sustained effects.

Participant Responsibilities:

Attend Weekly Sessions: Attend all scheduled mindfulness sessions. Daily Practice: Engage in daily mindfulness exercises and record their practice.

Keep a Diary: Maintain a diary or emotional response log of their emotional state, psychosocial experiences, and any adverse effects.

Outcome Measures:

Primary Outcome: Improvement in emotional intelligence as measured by SSEIT scores.

Secondary Outcomes:

Reduction in psychosocial distress as indicated by DASS scores. Improvement in trauma-related symptoms as measured by CATS. Monitoring and documentation of any adverse effects. Significance: This study aims to provide evidence on the effectiveness of mindfulness-based interventions in enhancing emotional intelligence and managing psychosocial challenges in adolescents with physical disabilities, potentially offering a valuable tool for improving their overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* The study would have the following inclusion criteria for participant recruitment.

  1. Adolescents with physical disability including:

     i. Orthopedic impairment ii. Traumatic brain injury iii. Sensory disability (vocally mute and partial visually impaired)
  2. Adolescents with physical disability in the age range 10-18
  3. Rural and urban residents
  4. Urdu, English and Punjabi speaking Participants who scored higher than cut off score on MAAS-A, DASS 21 SCS-SF, CATS and SSEIT in the phase I will be included in the phase II of the study i.e., Randomize control trail.

Exclusion Criteria:

* Exclusion Criteria The study would have the following inclusion criteria for participant recruitment.

  1. Adolescents under age 10 and above 18
  2. Adolescents who are not willing to participate or their guardians did not give permission will be excluded from the present study.
  3. Adolescents with physical disability such as:

     i. Fully visual impairment ii. Hearing impairment iii. Deaf-blindness iv. Severe psychiatric issue
  4. Also, participant with any chronic or comorbid disease will be excluded.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Emotional Intelligence | 8 weeks
  Improvement in emotional intelligence as measured by Schuttle Self Report Emotional Intelligence Test scores. The High Scores means more emotionally intelligent high Emotional Intelligence scores are typically above 123, average EI scores range from 90 to 122; and low EI scores are below 89 which means not that emotionally intelligent

CONTACTS AND LOCATIONS:
Locations (1):
- Aleeza Sohail, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No